CLINICAL TRIAL: NCT02070965
Title: Randomized Parallel Group Open-Label Multicenter Study to Assess the Potential for Adrenal Supp and Syst Drug Abs Following Multi Dosing With DFD-01 (Betamethasone Dipropionate) Spray 0.05% in Adol Subjects With Mod to Sev Plaque Psoriasis
Brief Title: DFD01 Spray vs Comp01 Lotion HPA Axis Suppression Study in Patients With Moderate to Severe Plaque Psoriasis
Acronym: BDS1307
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDS1307
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis

ARMS (3):
- DFD01 Spray Group 1 (Experimental): DFD01 Spray, bid, 28 days
  Interventions: Drug: DFD01 Spray
- Comp01 Lotion (Active Comparator): Comp01 Lotion, bid, 14 days
  Interventions: Drug: Comp01 Lotion
- DFD01 Spray Group 2 (Experimental): DFD01 Spray, bid, 14 days
  Interventions: Drug: DFD01 Spray

INTERVENTIONS:
Drug: DFD01 Spray
  Arms: DFD01 Spray Group 1; DFD01 Spray Group 2
Drug: Comp01 Lotion
  Arms: Comp01 Lotion

SUMMARY:
The purpose of this study is to evaluate the potential of DFD01 spray to suppress the HPA (hypothalamic-pituitary-adrenal) axis as compared to Comp01 lotion when applied twice daily for 15 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque psoriasis.
2. Subjects with psoriasis involving 20 to 50% BSA, not including the face, scalp, groin, axillae and other intertriginous areas.
3. Subjects must have an IGA grade of at least 3 (moderate) at the Baseline Visit
4. Subjects whose results from the screening ACTH stimulation test are considered normal (cortisol level >18 ug/dL at 30 minutes post stimulation) and show no other signs of abnormal HPA function or adrenal response. -

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
3. Have received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.
4. Use within 60 days prior to the Baseline Visit of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), or 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea)
5. Use within 30 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (salicylic acid, anthralin, coal tar, calcipotriene)2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy.
6. Use within 30 days prior to the Screening Visit of any product containing corticosteroids. Inhaled, intraocular, intranasal, etc. steroids are not allowed.
7. Subjects who have an abnormal sleep schedule or work at night.
8. Subjects with a known history of acute adrenal crisis, Addison's disease or decreased adrenal output, low pituitary function or pituitary tumors.
9. Subjects who have a history of an adverse reaction to cosyntropin injection or similar test reagents.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Encino Research Center T. Joseph Raoof MD, Inc., Encino, California
  - Redwood Dermatology Research, Santa Rosa, California
  - Bettencourt Skin Center, Henderson, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Suzanne Bruce and Associates, PA The Center for Skin Research Katy/Cinco Ranch, Katy, Texas

REFERENCES:
- [Derived] Sidgiddi S, Pakunlu RI, Allenby K. Efficacy, Safety, and Potency of Betamethasone Dipropionate Spray 0.05%: A Treatment for Adults with Mild-to-moderate Plaque Psoriasis. J Clin Aesthet Dermatol. 2018 Apr;11(4):14-22. Epub 2018 Apr 1. PMID 29657667

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD01 Spray Group 1: DFD01 Spray, bid, 28 days
  DFD01 Spray
- Comp01 Lotion: Comp01 Lotion, bid, 14 days
  Comp01 Lotion
- DFD01 Spray Group 2: DFD01 Spray, bid, 14 days
  DFD01 Spray
Period: Overall Study
Arm/Group | DFD01 Spray Group 1 | Comp01 Lotion | DFD01 Spray Group 2
Started | 27 | 23 | 25
Completed | 25 | 21 | 24
Not Completed | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Subject moved | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject signed informed consent and was randomized but was lost to follow up and, therefore, provided no baseline or post-baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD01 Spray Group 1 | Comp01 Lotion | DFD01 Spray Group 2 | Total
Number analyzed (Participants) | 27 | 22 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.99) | 45.4 (11.32) | 47.6 (13.71) | 46.7 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 9 | 21
  Male | 21 | 16 | 16 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 6
  White | 24 | 20 | 20 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 22 | 25 | 74
Percent Body Surface Area (BSA) involved [Mean (Standard Deviation); unit: Percent BSA affected] | 26.5 (8.61) | 26.8 (6.32) | 29.0 (11.04) | 27.4 (8.90)
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants]
  IGA 3 (Moderate) | 20 | 21 | 22 | 63
  IGA 4 (Severe/Very Severe) | 7 | 1 | 3 | 11
Normal Adrenal Corticotropic Hormone (ACTH) test [Count of Participants; unit: Participants] | 27 | 22 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With HPA Axis Suppression
Time Frame: Day 15
Population: Three subjects in the 28 day DFD01 Treatment Group, three subjects in the 14 day Comp01 Treatment Group, and one subject in the 14 day DFD01 Treatment Group did not have ACTH stimulation test results.
Measure: Count of Participants; unit: Participants
Arm/Group | DFD01 Spray Group 1 | Comp01 Lotion | DFD01 Spray Group 2
Number analyzed (Participants) | 24 | 20 | 24
Participants | 0 | 5 | 5

ADVERSE EVENTS:
Description: One subject signed informed consent and was randomized but was lost to follow up and, therefore, provided no baseline or post-baseline data.
Arm/Group | DFD01 Spray Group 1 | Comp01 Lotion | DFD01 Spray Group 2
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 2/27 | 6/22 | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray Group 1 (N=27) | Comp01 Lotion (N=22) | DFD01 Spray Group 2 (N=25)
HPA Axis Suppression (Endocrine disorders) | 0 (0) | 5 (5) | 5 (5)
Application Site Pruritus (General disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days